CLINICAL TRIAL: NCT03279042
Title: An Evaluation of the Efficacy of Conventional Corticotomy Versus Flapless Corticotomy in the En-Masse Retraction of Upper Anterior Teeth : A Randomized Controlled Trial
Brief Title: Effectiveness of Two Corticotomy Techniques in Retracting the Upper Anterior Teeth by Using Miniscrews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-04-2017
Record Dates: First submitted 2017-08-31; First posted 2017-09-12 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Class II Div 1 Malocclusion; Protrusion, Incisor
Keywords: En masse retraction; Corticotomy; Acceleration of tooth movement; Piezocision; Flapless corticotomy; Class II division 1 malocclusion; Protrusion of upper incisors; Sliding mechanics; mini-implant based anchorage; temporary anchorage devices
MeSH Terms: conditions — Malocclusion, Angle Class II; Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flapless corticotomy (Experimental): Flapless corticotomy will be conducted in this group of patients.
  Interventions: Procedure: Flapless corticotomy surgical intervention will be conducted
- Traditional corticotomy (Active Comparator): Traditional corticotomy will be performed in this group.
  Interventions: Procedure: Traditional corticotomy

INTERVENTIONS:
Procedure: Flapless corticotomy surgical intervention will be conducted — Piezocision will be used to perform the procedure
  Arms: Flapless corticotomy
Procedure: Traditional corticotomy — Here the surgery involves elevation of flaps and then conducting the surgical intervention using piezo-surgery cutting saws.
  Arms: Traditional corticotomy

SUMMARY:
This study aims to evaluate and compare the skeletal, dental and soft tissue changes, the levels of pain and discomfort and the effect on periodontal health and teeth vitality associated to traditional corticotomy and flapless corticotomy in the retraction of upper anterior teeth.

40 patients requiring extraction of maxillary first premolars and maximum anchorage to retract the upper anterior teeth will participate in the study. They will be divided randomly into two groups : flapless corticotomy (20 patients) and traditional corticotomy (20 patients). Pre-retraction, corticotomy will be performed in the maxillary anterior segment. The skeletal, dental and soft tissue changes will be performed using lateral cephalometric radiographs which will be obtained pretreatment, pre and post en-masse retraction of the anterior teeth and we will also use the dental casts to evaluate the dental changes.

DETAILED DESCRIPTION:
A corticotomy is cutting of the bone involves cortical bone only, leaving intact the medullary vessels and periosteum It offers an advantage to adult patients in reduction the orthodontic treatment time. The definition of traditional corticotomy is: elevating full-thickness periodontal flaps from a coronal approach, and vertical corticotomies are made between the teeth extending from 2-3 mm apical of the alveolar crest to 2 mm beyond the tooth apices and connected by a horizontal corticotomy; this process is done on both the labial and palatal aspects.

The definition of flapless corticotomy is: a minimally invasive version of corticotomy, using a piezotome in order to inflict bone injury. This technique entails labial and palatal interproximal piezoelectric microincisions into the cortical bone, without reflecting periodontal flaps.

Prior to enrollment of each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide a written informed consent.

Self-drilling titanium mini-implants (1.6mm diameter and 8mm length) will be used. they will be inserted between the maxillary second premolar and first molar at approximately 8-10mm above the archwires at the mucogingival junction and will be checked for primary stability (mechanical retention). Then the maxillary first premolar will be extracted. The maxillary arch will be levelled and aligned. The rectangular stainless steel archwires (0.019" × 0.025") with anterior 8mm height soldered hooks distal to the lateral incisors will be inserted.

The surgery will be carried out under local anesthesia. The traditional corticotomy will be handled by the same maxillofacial surgeon and the flapless corticotomy will be handled by the same orthodontist.

For traditional corticotomy, sulcular incisions the mesial aspect of one second premolar to the mesial surface of the contralateral second premolar will be placed, and full thickness flap will be elevated, 3 mm above the apical region of the tooth. piezoelectric under copious irrigation will be used for making vertical and horizontal cuts (only cortical surface). The vertical cuts will be between the dental roots in the interdental cortical surfaces ,stopping 2 mm short of the alveolar crest, occlusally. Horizontal cut will connect the vertical cuts 2 mm beyond root apex. These cuts will be performed from the mesial aspect of one second premolar to the mesial surface of the contralateral second premolar involving the anteriors. Similarly, a palatal flap incision will be raised immediately for doing the same vertical and horizontal cuts in the superficial surface of the palatal bone.

For the flapless corticotomy, The depth of gingival tissue will be determined through bone sounding using a periodontal probe. A scalpel will be used to make the incisions through the gingiva, 4mm below the interdental papilla to preserve the coronal attached gingiva. These vertical incisions will be placed from the mesial aspect of one second premolar to the mesial surface of the contralateral second premolar on the labial and palatal aspects of the maxilla through the gingiva and the underlying bone. A piezosurgery knife will be used to create the cortical alveolar incisions to a depth of 1 mm within the cortical bone.

Postoperatively, all patients will be advised to rinse with chlorhexidine mouthwash twice a day for one week. All patients will be contacted the day after the procedure to ensure no complications with surgery and will be followed up one month post-surgery to assess for signs of infection and ensure normal healing. We will assess patients' acceptance and the levels of pain and discomfort of traditional corticotomy and flapless corticotomy by asking all patients to fill out 4 questionnaires during the first month after the surgical procedure using a VAS.

The surgical procedure will be performed and (250-300) g force will be applied on each side (3-4 days) after corticotomy using two NiTi springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction. The force level will be measured every 2 weeks after the corticotomy . Retraction will be stopped when a class I canine relationship will be achieved and a good incisor relationship will be obtained.

Periodontal health will be assessed at the beginning of orthodontic treatment, before and after corticotomy by evaluating the following parameters: plaque index, gingival index, bleeding index, and gingival recession.

Dental casts will be used for the quantification of the anteroposterior movement of the anterior teeth and the first molars every 30 days until class I canine relationship will be achieved and a good incisor relationship will be obtained.

To evaluate the movement of the anterior teeth: we will project the canine cusp on the median line and measure the distance from this point to the projected position of a distinct medial ruga point.

To evaluate the movement of the first molars: we will project the mesial contact point of the first molar on the median line and measure the distance from this point to the projected position of a distinct medial ruga point. These measurements will be made with sliding calipers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with permanent occlusion at age 18-30 years.
* Comprehensive medical and dental history ruling out any systemic disease
* Not under any systemic medication.
* No previous orthodontic treatment
* Patients with satisfactory periodontal health and Good oral hygiene
* Need to orthodontic treatment with fixed appliances
* No congenitally missing teeth except third molars in the maxillary arch
* Mild or no anterior crowding in maxillary arch.
* Maximum anchorage, with 75% to 100% of space closure of retraction of anterior segment in maxillary arch.
* Therapeutic extraction of maxillary first premolars required.
* Patients with class Ⅱ division 1 (ANB angle ≤7 degrees) with severe overjet (5-10 mm)
* Maximum retraction of the anterior teeth was desired.

Exclusion Criteria:

* Patients with previous orthodontic treatment.
* Patients with severe skeletal dysplasia in all three dimensions.
* Patients suffer from systemic diseases or syndromes
* Patients on medication for systemic disorders, pregnancy or steroid therapy.
* Patients showing any signs of active periodontal disease
* Patients with severe crowding (≥ 3.5 mm) in maxillary arch
* Patients with missing or extracted teeth in maxillary arch except third molar.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Duration of en-masse retraction of anterior teeth | The months required to compete the retraction procedure will be recorded. Completion of this procedure is expected to be occur within six months in the experimental group and eight months in the control group.
  Assessment will be performed by calculating the months required to achieve complete retraction of the upper anterior teeth (six teeth) through clinical examination.
Rate of retraction | The calculation of the rate of retraction will be done once the retraction procedures has finished. Completion of this procedure is expected to occur within 6 months in the experimental group and 8 months in the control group.
  Assessment will be performed on study models. The amount of distance being retracted in millimeters will be divided by the duration of retraction in weeks to give an estimation of the retraction rate.
Change in Incisors' positions | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  Amount of distance being traveled by the retracted anterior teeth is going to be measured on study models taken at monthly intervals until the end of the retraction phase.
Change in Molars' positions | T0: 1 day before the beginning of retraction. T1: after 1 month (m) of retraction. T2: after 2 m of retraction. T3: after 3 m. T4: after 4 m. T5: at the end of retraction (expected to be within 6 m in the exp. group and 8 m in the control group)
  Amount of distance being traveled by the first molars and is going to be measured on study models taken at monthly intervals until the end of the retraction phase.
Change in the SNA angle | The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SNB angle | The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the ANB angle | The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SN.GoMe angle | The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the amount of backward rotation of the lower jaw in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the MM angle | The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.

SECONDARY OUTCOMES:
Change in the levels of pain and discomfort | Levels of pain will be assessed at : 24 hours following the surgical intervention (T1), one week (T2) , two weeks (T3) and four weeks (T4) following the surgical intervention
  Assessment will be performed using questionnaires via visual analog scales (VAS)
Change in the Plaque index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The plaque index will be used to assess the status of the oral hygiene in these patients.
Change in the Gingival index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The Gingival index will be used to assess the status of the gingival tissues around the teeth.
Change in the Bleeding index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The plaque index will be used to assess the status of periodontal tissues and the amount of congestion in the gingival margins around the anterior teeth.
Gingival Recession | Two measurements are required for this calculation: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  This will be measured in millimeters from the cement-enamel junction to the level of the gingival margin around the six anterior teeth.
Change in Tooth Vitality | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  Tooth vitality will be evaluated for each tooth of the six anterior teeth using Ethyl Chloride applied by a cotton roll.

CONTACTS AND LOCATIONS:
Overall Officials: Hanin Nizar Khlef, DDS, Principal Investigator — MSc student, Department of Orthodontics, University of Damascus Dental School, Syria; Mohammad Y Hajeer, DDS MSc Phd, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Syria; Omar Hashmeh, DDS MSc PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192
- [Background] Seo KW, Kwon SY, Kim KA, Park KH, Kim SH, Ahn HW, Nelson G. Displacement pattern of the anterior segment using antero-posterior lingual retractor combined with a palatal plate. Korean J Orthod. 2015 Nov;45(6):289-98. doi: 10.4041/kjod.2015.45.6.289. Epub 2015 Nov 20. PMID 26629475
- [Background] Lee J, Miyazawa K, Tabuchi M, Sato T, Kawaguchi M, Goto S. Effectiveness of en-masse retraction using midpalatal miniscrews and a modified transpalatal arch: Treatment duration and dentoskeletal changes. Korean J Orthod. 2014 Mar;44(2):88-95. doi: 10.4041/kjod.2014.44.2.88. Epub 2014 Mar 19. PMID 24696825
- [Background] Krishnan P, Shetty S, Husain A. An adjunctive minor surgical procedure for increased rate of retraction. J Pharm Bioallied Sci. 2013 Jun;5(Suppl 1):S39-42. doi: 10.4103/0975-7406.113293. PMID 23946574
- [Background] Jee JH, Ahn HW, Seo KW, Kim SH, Kook YA, Chung KR, Nelson G. En-masse retraction with a preformed nickel-titanium and stainless steel archwire assembly and temporary skeletal anchorage devices without posterior bonding. Korean J Orthod. 2014 Sep;44(5):236-45. doi: 10.4041/kjod.2014.44.5.236. Epub 2014 Sep 25. PMID 25309863
- [Background] Sakthi SV, Vikraman B, Shobana VR, Iyer SK, Krishnaswamy NR. Corticotomy-assisted retraction: an outcome assessment. Indian J Dent Res. 2014 Nov-Dec;25(6):748-54. doi: 10.4103/0970-9290.152191. PMID 25728107
- [Background] Bhattacharya P, Bhattacharya H, Anjum A, Bhandari R, Agarwal DK, Gupta A, Ansar J. Assessment of Corticotomy Facilitated Tooth Movement and Changes in Alveolar Bone Thickness - A CT Scan Study. J Clin Diagn Res. 2014 Oct;8(10):ZC26-30. doi: 10.7860/JCDR/2014/9448.4954. Epub 2014 Oct 20. PMID 25478442
- [Background] Chung KR, Mitsugi M, Lee BS, Kanno T, Lee W, Kim SH. Speedy surgical orthodontic treatment with skeletal anchorage in adults--sagittal correction and open bite correction. J Oral Maxillofac Surg. 2009 Oct;67(10):2130-48. doi: 10.1016/j.joms.2009.07.002. PMID 19761907
- [Derived] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O, Youssef N, Mahaini L. The effectiveness of traditional corticotomy vs flapless corticotomy in miniscrew-supported en-masse retraction of maxillary anterior teeth in patients with Class II Division 1 malocclusion: A single-centered, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2020 Dec;158(6):e111-e120. doi: 10.1016/j.ajodo.2020.08.008. Epub 2020 Nov 4. PMID 33158633